CLINICAL TRIAL: NCT04138719
Title: Clinical Study of Nab-paclitaxel Plus Carboplatin Versus Nab-paclitaxel Plus Epirubicin in the Neoadjuvant Therapy for Breast Cancer
Brief Title: Nab-paclitaxel Plus Carboplatin Versus Nab-paclitaxel Plus Epirubicin in the Neoadjuvant Therapy for Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Collaborators: Beijing 302 Hospital (Other); CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Cuizhi GENG, M.D., Hebei Medical University Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-KAL-BC-11
Record Dates: First submitted 2019-10-23; First posted 2019-10-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Triple-negative Breast Cancer; Nab-paclitaxel
Keywords: Triple-negative Breast Cancer; Nab-paclitaxel; Carboplatin; Epirubicin
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Carboplatin; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nab-paclitaxel + Carboplatin (Experimental): nab-paclitaxel given IV at 125 mg/m^2 on days 1, 8 and carboplatin given IV at AUC 5 on days 1 every 21 days x 6 cycles；
  Interventions: Drug: Nab-paclitaxel + Carboplatin
- Nab-paclitaxel + Epirubicin (Active Comparator): nab-paclitaxel given IV at 125 mg/m^2 on days 1, 8 and epirubicin given IV at 75 mg/m^2 on days 1 every 21 days x 6 cycles；
  Interventions: Drug: Nab-paclitaxel + Epirubicin

INTERVENTIONS:
Drug: Nab-paclitaxel + Carboplatin — nab-paclitaxel given IV at 125 mg/m^2 on days 1, 8 and carboplatin given IV at AUC 5 on days 1 every 21 days x 6 cycles;
  Arms: Nab-paclitaxel + Carboplatin
Drug: Nab-paclitaxel + Epirubicin — nab-paclitaxel given IV at 125 mg/m^2 on days 1, 8 and epirubicin given IV at 75 mg/m^2 on days 1 every 21 days x 6 cycles；
  Arms: Nab-paclitaxel + Epirubicin

SUMMARY:
This is a multicenter, open, randomized, comparison study. Triple-negative breast cancer (TNBC) is a term applied to breast cancer cases that have <1% expression of the estrogen receptor (ER) and the progesterone receptor (PR) and do not over express HER2.

Neoadjuvant therapy is often used to reduce the size of tumors, especially in locally advanced tumors. The purpose of this therapy is to make part of patients operable and to facilitate breast-conserving surgery.

The purpose of this study is to assess the efficacy and safety of the following two proposals: nab-paclitaxel plus carboplatin versus nab-paclitaxel plus epirubicin, in order to provide support for rational clinical application.

The total number of patients to be included in this study is 520 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 to 70 years old;
2. Histologically confirmed primary invasive breast cancer;
3. Histologically confirmed triple negative breast cancer;
4. Patients who planned to accept preoperative neoadjuvant therapy and had a mass larger than 2 cm.
5. Blood specimens and 5 sections of tumor tissue at baseline, blood specimens at surgery can be obtained.
6. Have at least one measurable lesion as per the RECIST criteria (version 1.1);
7. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to one;
8. LVEF≥55%；
9. Bone marrow function：neutrophils (≥1.5×10^9/L), platelets (≥100×10^9/L), hemoglobin (≥90 g/L);
10. Renal and hepatic function: Serum creatinine≤ 1.5×institutional upper limit of normal (ULN); AST and ALT ≤ 2.5 × ULN; Total bilirubin≤1.5×ULN, or patients with Gilbert's syndrome ≤ 2.5 × ULN;
11. Patients had good compliance with the planned treatment, understood the research process and written informed consent.

Exclusion Criteria:

1. Previous treatment with any cytotoxic chemotherapy, endocrine therapy, biotherapy or radiotherapy;
2. Patients with heart disease above grade II (including grade II) identified by New York Heart Association (NYHA) scores;
3. Patients with severe systemic infection or other serious diseases;
4. Patients allergic to or intolerant of chemotherapeutic drugs or their adjuvants;
5. Patients with other malignant tumors in the past five years, except for cured cervical carcinoma in situ and non-melanoma skin cancer;
6. Pregnancy or lactation, as well as reproductive age patients who refused to take appropriate contraceptive measures in the trial;
7. Participation in any trial drug treatment or another interventional clinical trial 30 days before first dose was given;
8. The researchers considered the patients who were not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 520 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
pCR (pathological complete response) | 3 years
  No residual infiltrating cancer cells were found in surgical specimens of breast and axillary lymph nodes; residual cancer cells in situ in surgical specimens can also be considered to achieve pCR

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 years
Disease free survival（DFS） | 3 years
Adverse events (AE) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, M.D., Study Chair — Beijing 302 Hospital; Cuizhi Geng, M.D., Study Chair — Hebei Medical University Fourth Hospital
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No